CLINICAL TRIAL: NCT04746768
Title: Impact of Exercise and Nutritional Support on the Frailty Syndrome of Eldery Patients in Phase of Post-cancer Treatment
Brief Title: Frailty Syndrome of Post-cancer Treatment Eldery Patients
Acronym: PANACEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC19.144
Record Dates: First submitted 2020-11-26; First posted 2021-02-10 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-02

CONDITIONS: Frailty Syndrome; Exercise; Nutritional Support; Cancer
MeSH Terms: conditions — Frailty; Motor Activity; Neoplasms | interventions — Exercise; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise and nutritional support (Experimental): exercise and nutritional support program during an active support phase (0 to 6 months) followed by an empowerment phase (from 6 to 12 months)
  Interventions: Combination Product: exercise and nutritional support

INTERVENTIONS:
Combination Product: exercise and nutritional support — exercise and nutritional support program during an active support phase (0 to 6 months) followed by an empowerment phase (from 6 to 12 months)

SUMMARY:
Decrease the prevalence of frailty syndrome in individuals with complete response of cancer.

ELIGIBILITY:
Inclusion Criteria:

* in complete remission from cancer (all type of cancer)
* have a frailty syndrome (positive GFST score)
* ability to provide signed informed consent
* be affiliated with social security or beneficiary of such a scheme

Exclusion Criteria:

* patient with active cancer or any other pathology affecting the prognosis at 5 years
* currently participating or having participated in the month preceding inclusion in another interventional clinical research that may impact the study. This impact is left to the investigator discretion
* subjects referred to articles L1121-5 to L1121-8 of CSP (corresponds to all protected persons: person deprived of liberty by judicial or administrative decision, person subject to legal protection measure)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change of the prevalence of frailty syndrome in individuals with complete response of cancer | 0, 6 and 12 months
  evolution of individual frailty during a multimodal intervention (physical and nutritional activity) according to the Fried's criteria

SECONDARY OUTCOMES:
evaluation of predicitive variables of frailty syndrome reversion | Month 0, 6 and 12
  The criterion determining the frail status is the Fried score classified into 3 categories: not frail; pre-frail; frail. A change from frail to pre-frail or to not frail will be considered as an improvement. Measurements of the Frailty score and other markers on nutrition and APA will be carried out at month 0 (basic measurements), then measured at month 6 (end of APA and nutritionist support) and at month12 (6 months after empowerment). All of health markers collected during the basic assessment, changes in parameters (month 6) and compliance with APA and nutrition support (from Month 1 to Month 6 then between Month 6 and Month 12) will be tested as variables potentially predictive of an improvement in the frailty syndrome.
Correlations between physical performance and frailty syndrome and their evolutions | Month 0, 6 and 12
  measurement of VO2peak + ventilatory thresholds measured in a stress test, muscle strength/endurance (number of chair raises for 30 seconds), walking speed (10-meter walking test, 6-minute walk test), balance (Tinette score), coordination (functional mobility test), cardio-respiratory endurance (heart rate measurement in relation to pedaling power)
Change from baseline nutritional status during nutritionist support (month 3 and 6) and at the end of empowerment (month 12) | Month 0, 3, 6 and 12
  nutritional parameters measured at each time frame for weight, VAS appetite score, MNA score, nutritional calculation (food survey and self-questionnaire), bio impedancemetry and biomarkers of nutrition (levels of albumin, prealbumin, C reactive protein, CBC, liver and kidney function)
Measure adherence to APA interventions and exercise practices | between month 1 to 6 and between month 6 to 12
  Adherence to APA support program throughout the study will be evaluated by measurements and sum of multiple parameters: number of sessions recorded on the heart rate monitor, average energy expenditure (in kcal) measured by the heart rate monitor,number of sets of exercises performed relative to the number of exercises recommended for muscle strengthening recorded in the patient notebook, CESS scale to assess beliefs about cancer patients and physical activity
Estimation of adherence to nutritional interventions | Month 6 and 12
  comparison between active support phase and empowerment phase with food self-questionnaire
Measure the durability of long-term activities | Month 6 and 12
  number of monthly patient connections to heart rate monitor; evaluation of the completion of patient notebook
Measure health related quality of life on mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression | Month 0, 6 and 12
  Assessment of quality of life with EQ-5D questionnaire by comparison to the basal state (M0).
Sociological study on motivation: evaluation of the perception and experience of treating patients | Month 6 and 12
  a series of qualitative interviews with a panel of 15 patients, during 2 interview sessions: 1 after support phase and 1 at the end of autonomy phase. Interview will collect past/current socio-professional life, socialization in physical activity and nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Gavazzi, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble, Grenoble, France